CLINICAL TRIAL: NCT06279507
Title: The Efficacy of Hyaluronic Acid Injection as an Adjunctive Treatment After Intraarticular Low-dose Glucocorticoid Injection for Symptomatic Knee Osteoarthritis: A Multicenter Randomized, Controlled, Double-blinded Study
Brief Title: Efficacy of Hyaluronic Acid Injection in Knee Osteoarthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Chulalongkorn University (Other); Khon Kaen University (Other); Police General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMK-00007
Record Dates: First submitted 2023-10-07; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis; Pain, Joint; Stiffness of Knee, Not Elsewhere Classified; Quality of Life
Keywords: Hyaluronic acid; Adjunctive treatment
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia | interventions — Hyaluronic Acid; Saline Solution; Sodium Chloride; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: The participants would be allocated into one treatment group;
  * Intervention group : Hyaluronic acid injection
  * Placebo group : Normal saline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not know what treatment they receive. Co-investigators will not know what the participants are injected. Outcome assessor will not know which treatment participant receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid (Active Comparator): Hyaluronic acid, Ostenil Plus, 2 mL (40 mg) will be injected once afer 2-4 week of glucocorticoid injection
  Interventions: Drug: Sodium Hyaluronate; Drug: Triamcinolone Acetonide 10mg/mL
- Normal saline (Placebo Comparator): Two-millilitres of normal saline will be injected once after 2-4 weeks of glucocorticoid injection
  Interventions: Drug: Normal Saline; Drug: Triamcinolone Acetonide 10mg/mL

INTERVENTIONS:
Drug: Sodium Hyaluronate — Sodium hyaluronate 2% (40 mg/2 mL), with molecular weight of 1-2 million dalton Other active ingredient : Mannitol 0.5% Preparation : Pre-filled syringe
  Other Names: Ostenil Plus
  Arms: Hyaluronic acid
Drug: Normal Saline — 0.9% sodium chloride 2 mL prepared in plastic syringe
  Other Names: 0.9% sodium chloride
  Arms: Normal saline
Drug: Triamcinolone Acetonide 10mg/mL — 10 mg of triamcinolone acetonide will be injected to all participants before the specified intervention

SUMMARY:
The aim of this clinical trial study is to compare the efficacy of Hyaluronic injection in patients with symptomatic knee osteoarthritis. The main questions it aims to answer are:

* Is Hyaluronic acid injection improve pain symptom, joint stiffness, and joint function in patients with knee osteoarthritis
* Is Hyaluronic acid injection improve knee performance status and health-related quality of life in patients with knee osteoarthritis

Participants will be allocated to receive one treatments; either Hyaluronic acid or normal saline injections after receiving glucocorticoid injection.

Researchers will compare the Hyaluronic acid with normal saline injection to see if the former show superior effect in terms of pain, joint stiffness, function, as well as health-related quality of life comparing with placebo.

DETAILED DESCRIPTION:
Participants who had been diagnosed with knee osteoarthritis according to American College of Rheumatology (ACR) criteria will be enrolled in this study. After the participants receive the information and consent to participate in this study, they will be examined their affected knee by the co-researchers. Ten-milligrams of Triamcinolone will be injected intra-articular into knee joint.

Two-to-four weeks later, the participants will be evaluated for knee pain, stiffness, function and quality of life, as well as knee performance status. Participants whose their knee joint absence of effusion will be allocated in to one treatment group; either Hyaluronic acid or normal saline. After injection, participants will be scheduled for the follow-up visit in 12 and 24 weeks later. In each follow-up visit, they will be evaluated for joint pain, stiffness, function and quality of life, as well as analgesic use and adverse reaction form treatment.

ELIGIBILITY:
Inclusion Criteria:

* All participants who had been diagnosed as knee osteoarthritis according to ACR criteria with symptom of knee pain
* Pain visual analog scare of 4 or higher

Exclusion Criteria: Participants who have

* Cognitive impairment
* History of aller to Hyaluronic acid or its component
* History of knee arthropathy
* Concomitant with inflammatory arthritis
* Serious comorbidities or bedridden status
* Current pregnancy or lactation
* Currently use of symptomatic slow acting drugs for osteoarthritis (SYSADOA)
* Communication problem

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain outcome measurement | 12 and 24 weeks after injection
  The comparison between Hyaluronic acid and normal saline injection in the change of joint pain after the injection, by using visual analog scale and pain domain assessment in Western Ontario and McMaster University (WOMAC) scale (scale 0-10, which higher scale reflects worse symptom)
Joint stiffness and function measurement | 12 and 24 weeks after injection
  The comparison between Hyaluronic acid and normal saline injection in the change of joint stiffness and function after the injection, by using WOMAC scale (scale 0-10, which higher scale reflects worse symptom or function)
Overall symptom assessment | 12 and 24 weeks after injection
  The comparison between Hyaluronic acid and normal saline injection in the change of overall symptom after the injection, by using patient's global assessment (scale 0-10, which higher scale reflects worse condition)

SECONDARY OUTCOMES:
Knee performance evaluation | 12 and 24 weeks after injection
  The comparison between Hyaluronic acid and normal saline injection in the change of knee performance status after the injection, assessed by Time Up and Go test
Quality of life assessment | 12 and 24 weeks after injection
  The comparison between Hyaluronic acid and normal saline injection in the change of health-related quality of life assessed by EuroQol group - 5 Dimensions - 5 Levels (EQ-5D-5L) tool (scale 0-100, which higher scale reflects better health)

CONTACTS AND LOCATIONS:
Overall Officials: Nis Okuma, Medical, Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No